CLINICAL TRIAL: NCT07221097
Title: Prospective Clinical Evaluation of the BioFire Emerging Coronavirus Panel - Sponsor's Protocol
Brief Title: Prospective Clinical Evaluation of the BioFire Emerging Coronavirus Panel for the Detection of COVID-19 and Other Coronaviruses
Status: Recruiting | Type: Observational
Sponsor: BioFire Defense LLC (Industry)
Collaborators: Children's Hospital Los Angeles (Other); George Washington University (Other); Wake Forest University Health Sciences (Other); Tampa General Hospital (Other); The University of Texas Medical Branch, Galveston (Other); Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: DF-SDY-034538; 75A50122C00073 (Other Grant/Funding Number: Biomedical Advanced Research and Development Authority)
Record Dates: First submitted 2025-10-22; First posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Coronavirus; Respiratory Infection; COVID
Keywords: in vitro diagnostic; pandemic preparedness; medical device; molecular diagnostic; coronavirus
MeSH Terms: conditions — Coronavirus Infections; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nasopharyngeal swabs (NPS) eluted in transport medium
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Suspected respiratory infection: NPS specimens leftover from SOC testing for a suspected respiratory infection as determined by a health care provider
  Interventions: Device: Investigational IVD for coronaviruses

INTERVENTIONS:
Device: Investigational IVD for coronaviruses — Device testing on prospectively collected specimens leftover from standard of care for IVD validation only; results will not influence patient care/management.
  Other Names: BIOFIRE ECoV Panel

SUMMARY:
The Biomedical Advanced Research and Development Authority (BARDA) has contracted BioFire Defense (BFDf) to develop the BioFire Emerging Coronavirus (ECoV) Panel, a nucleic acid test capable of detecting coronaviruses from nasopharyngeal swab (NPS) in transport medium.

This study aims to evaluate the diagnostic accuracy of the assays comprising the BioFire ECoV Panel. It is hypothesized that the BioFire ECoV Panel assays will be highly sensitive and specific for the detection of the coronaviruses included on the panel.

DETAILED DESCRIPTION:
The primary objective of this observational, non-interventional study is to evaluate the diagnostic accuracy of the assays comprising the BioFire ECoV Panel when used to test NPS obtained from individuals with signs and/or symptoms of respiratory infection. Multiple geographically distinct clinical sites in the U.S. will participate in testing. Enrollment will consist of residual, coded NPS specimens leftover from standard of care testing for a suspected respiratory infection as determined by a health care provider. Concordance between the BioFire ECoV Panel assays and comparator methods will be measured using positive and negative percent agreement (PPA and NPA).

ELIGIBILITY:
Inclusion Criteria:

* Specimen is residual NPS in transport medium (VTM or UTM) left over from standard of care testing under clinician order for respiratory pathogen analysis.
* Specimen has been held at room temperature for less than or equal to 4 hours or 4°C for less than or equal to 72 hours before enrollment.
* At least 1.7 mL of specimen is remaining after standard of care testing and available for use in the study

Exclusion Criteria:

* Specimen is unable to be tested within the defined storage parameters
* Insufficient specimen volume for testing
* Transport medium type is unknown

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients suspected of a respiratory infection by their healthcare provider
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Device Performance | Through study completion; September 2025-August 2026
  Positive Percent Agreement and Negative Percent Agreement for Panel Targets

CONTACTS AND LOCATIONS:
Overall Officials: Brittany C Collins, PhD, Principal Investigator — BioFire Defense LLC
Locations (6):
- United States (6):
  - Children's Hospital Los Angeles, Los Angeles, California
  - George Washington University, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://medicalcountermeasures.gov/barda/barda-covid-19-response/covid-19-portfolio